CLINICAL TRIAL: NCT03600584
Title: Modified One-layer Duct-to-mucosa Versus Invagination for Pancreaticojejunostomy After Pancreaticoduodenectomy
Brief Title: Modified Duct-to-mucosa Pancreaticojejunostomy After Pancreaticoduodenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yi Miao, Prof., Director of Pancreas Center, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JSPH-PC-201801
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Pancreatic Fistula
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-layer duct-to-mucosa Group (Experimental): Modified one-layer duct-to-mucosa pancreaticojejunostomy is used after pancreaticoduodenectomy.
  Interventions: Procedure: Modified one-layer duct-to-mucosa Pancreaticojejunostomy
- Invagination Group (Active Comparator): Invagination pancreaticojejunostomy is used after pancreaticoduodenectomy.
  Interventions: Procedure: Invagination pancreaticojejunostomy

INTERVENTIONS:
Procedure: Modified one-layer duct-to-mucosa Pancreaticojejunostomy — After the completion of the preparation of the remnant pancreas for reconstruction was performed. Modified one-layer duct-to-mucosa Pancreaticojejunostomy was performed.
  Arms: One-layer duct-to-mucosa Group
Procedure: Invagination pancreaticojejunostomy — After the completion of the preparation of the remnant pancreas for reconstruction was performed. Invagination Pancreaticojejunostomy was performed.
  Arms: Invagination Group

SUMMARY:
The aim of this study is to compare surgical outcomes of modified One-layer duct-to-mucosa versus invagination pancreaticojejunostomy after pancreatoduodenectomy

DETAILED DESCRIPTION:
Duct-to-mucosa and invagination pancreaticojejunostomy are two most commonly used anastomotic techniques after pancreaticoduodenectomy, with comparable incidence rate of pancreatic fistula (PF). We modified the conventional two-layer duct-to-mucosa PJ into one-layer PJ. The aim of this study is to examine if the investigator's modified duct-to-mucosa PJ can reduce PF after PD when compared to invagination PJ.

This trial is a single-center, randomized, controlled, patient- and observer- blinded study, whose primary aim is to assess whether a modified duct-to-mucosa PJ (trial group) is superior to an invagination PJ (control group), in terms of clinically relevant PF and other complications. A total of 380 patients, who are to undergo elective PD, will be recruited and randomized intraoperatively into either of the two groups. The primary efficacy endpoint is the incident rate of clinically relevant PF. Secondary outcome measures are: entry into adjuvant therapy, mortality, surgical complications, non-surgical complications, hospital stay. Patients will be followed up for 3 months. Statistical analysis will be based on the intention-to-treat population. The duration of the entire trial is estimated to be two years.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed consent obtained；
* Both sexes between 18 and 80 years old；
* Patients scheduled to elective open pancreaticoduodenectomy.

Exclusion Criteria:

* Patients with ASA score >=4;
* Patients who had a previous pancreatic operation;
* Patients with an immunodeficiency;
* Patients who underwent an emergency operation;
* Pregnant patients；
* Patients who was found that pancreaticoduodenectomy was not suitable。

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Rate of clinically relevant postoperative pancreatic fistula (POPF) | Up to 60 days after Surgery
  As defined by International Study Group on Pancreatic Fistula, a clinically relevant postoperative pancreatic fistula is now redefined as a drain output of any measurable volume of fluid with an amylase level >3 times the upper limit of institutional normal serum amylase activity, associated with a clinically relevant development/condition related directly to the postoperative pancreatic fistula.

SECONDARY OUTCOMES:
Anastomosis time | intraoperatively
  Time from the beginning to the end of the pancreatic reconstruction
Delayed gastric emptying | Up to 60 day after Surgery
  The International Study Group for Pancreatic Surgery definition and classification of delayed gastric emptying were applied. Briefly, grade A, unable to tolerate solid oral intake by POD 7 and usually no vomiting; grade B, unable to tolerate solid oral intake by POD 14 with/without vomiting: and grade C, unable to tolerate solid oral intake by POD 21 with/without vomiting.
post-pancreatectomy hemorrhage (PPH) | Up to 60 days after Surgery
  The 2017 International Study Group for Pancreatic Surgery definition and classification of PPH were applied.
Chyle leak | Up to 60 days after Surgery
  The 2017 International Study Group for Pancreatic Surgery definition and classification of chyle leak were applied.
Overall Morbidity | Up to 60 days after Surgery
  Any complications that occur postoperatively. The severity of complications was graded according to the Clavien-Dindo classification.
Mortality | Up to 90 days after Surgery
  Patient death that occurs postoperatively
Reoperation rate | Up to 90 days after Surgery
  Patients who needs a surgical re-operation for any reasons during the postoperative hosptial stay. Reasons and times of reoperation are recorded.
Readmission rate | Up to 60 days after Surgery
  Patients that readmitted into hospital for reasons that related to complications of last pancreatic surgery.
Duration of postoperative hospital stay | Up to 90 days after Surgery
  Time from day of operation to day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Miao, Prof., Study Director — Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wei J, Liu X, Wu J, Xu W, Zhou J, Lu Z, Chen J, Guo F, Gao W, Li Q, Jiang K, Dai C, Miao Y. Modified One-layer Duct-to-mucosa Pancreaticojejunostomy Reduces Pancreatic Fistula After Pancreaticoduodenectomy. Int Surg. 2015 Jun 3. doi: 10.9738/INTSURG-D-15-00094.1. Online ahead of print. PMID 26037262
- [Derived] Hai H, Li Z, Zhang Z, Cheng Y, Liu Z, Gong J, Deng Y. Duct-to-mucosa versus other types of pancreaticojejunostomy for the prevention of postoperative pancreatic fistula following pancreaticoduodenectomy. Cochrane Database Syst Rev. 2022 Mar 15;3(3):CD013462. doi: 10.1002/14651858.CD013462.pub2. PMID 35289922